CLINICAL TRIAL: NCT05095571
Title: A Randomized Placebo-controlled Trial of Nicotinamide/Pterostilbene Supplement in ALS: The NO-ALS Study. Extension Protocol
Brief Title: A Trial of Nicotinamide/Pterostilbene Supplement in ALS: The NO-ALS Extension Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Elysium Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 266376
Record Dates: First submitted 2021-10-04; First posted 2021-10-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — nicotinamide-beta-riboside; Pterocarpus marsupium

STUDY DESIGN:
Intervention Model Description: The study is a multicenter open label study as a follow up of the NO-ALS trial. Newly diagnosed ALS cases were included in the study arm 1. Earlier ALS cases were included in study arm 2 to allow patients with earlier ALS to participate in the study as the treatment options outside the study were limited. The NO-ALS study will be stopped when we reach 180 patients in the group with newly diagnosed ALS cases (arm 1). This is the follow up study for patients completing 1 year follow up in the NO-ALS study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NO-ALS Extension Study High Dose EH301 (Other)
  Interventions: Dietary Supplement: EH301 (Nicotinamide Riboside/Pterostilbene)

INTERVENTIONS:
Dietary Supplement: EH301 (Nicotinamide Riboside/Pterostilbene) — For this study EH301 is defined as Investigational Product(s) (IP). The ALS extension study is an open label study with active treatment of all patients thet have passed through the NO-ALS trial.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a serious rapidly progressive disease of the nervous system. The mean survival from the time of diagnosis is 2.5 years. Apart from Riluzole, there is no effective treatment. Care of advanced ALS will have a cost of 4-8 million NOK (Norwegian kroner) per year.

Research i.a. from the investigators department has shown that increased activity in histone deacetylation enzymes (sirtuins) together with increased access to Nicotinamide Adenine Dinucleotide (NAD) can delay disease progression. Nicotinamide riboside (NR) can increase cells' access to NAD and Pterostilbene will stimulate sirtuins.

The investigators want to study whether combination therapy with NR and Pterostilbene can inhibit neurodegeneration in ALS and thereby delay disease development, increase survival and improve quality of life in ALS.

In the NO-ALS extension study the investigators will follow the patients who completed the original NO-ALS study. Objectives are to evaluate adverse events and give patients possibility of compassionate use, and secondarily to see if the combination of NR and pterostilbene (EH301) will decrease progression of motor symptoms and loss of vital capacity, and increase survival time in patients with ALS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfilled the criteria for the NO-ALS study and have completed the study will be proposed inclusion in the NO-ALS extension study protocol. Patients from both arm 1 and arm 2 in the NO-ALS study will be allowed inclusion in the prolongation study

Exclusion Criteria:

Individuals will be excluded if any of the following exclusion criteria apply:

* Dementia, fronto temporal dementia (FTD) or other neurodegenerative disorder interfering with compliance.
* Metabolic, neoplastic, or other physically or mentally debilitating disorder.
* Patients who become tracheostomized as part of the treatment of ALS.
* Patients with short expected survival at the discretion of the investigator. Such cases cannot be expected to follow protocol procedures.
* Use of Vit B3 or blue berry extracts outside the study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through study completion, 1 year
  Studies of adverse events including changes in lab parameters induced by high dose oral NR/pterostilbene.

SECONDARY OUTCOMES:
Disease progression as assessed by Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) | Determined after 12 months of follow-up.
  ALSFRS-R is a validated rating instrument for monitoring the progression of disability in patients with ALS. The minimum score is 0 and the maximum score is 48, the higher score the more function is retained.
Change in vital capacity | Determined after 12 months of follow-up.
  Vital capacity measured by spirometry.

OTHER OUTCOMES:
Overall survival | Determined after 12 months of follow-up.
  Defined as how many are alive or not requiring continuous respiratory ventilation life support.

CONTACTS AND LOCATIONS:
Overall Officials: Ole-Bjørn Tysnes, Principal Investigator — Haukeland University Hospital
Locations (17):
- Norway (17):
  - Haukeland University Hospital, Bergen
  - Nordlandssykehuset HF, Bodø
  - Vestre Viken HF, Drammen
  - Helse Førde HF, Førde
  - Helse Fonna HF, Haugesund
  - Sørlandet sykehus, Kristiansand
  - Sykehuset Innlandet HF, Lillehammer
  - Akershus University Hospital, Lørenskog
  - Helse Møre og Romsdal, Molde
  - Helse Nord-Trøndelag HF, Namsos
  - Oslo Univerity Hospital, Oslo
  - Sykehuset Østfold HF, Sarpsborg
  - Sykehuset i Telemark HF, Skien
  - Stavanger University Hospital, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø
  - St. Olavs Hospital HF, Trondheim
  - Sykehuset i Vestfold HF, Tønsberg